CLINICAL TRIAL: NCT02700386
Title: Hypofractionated, Comprehensive Radiation Therapy for Node-Positive Breast Cancer
Brief Title: Shorter Course Radiation for the Treatment of Breast Cancer That Has Spread to Lymph Nodes
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-1329.cc
Record Dates: First submitted 2016-02-22; First posted 2016-03-07 (Estimated); Results first posted 2025-04-20 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
Keywords: Breast; Cancer; Hypofractionated; Node-Positive Breast Cancer; Radiation Therapy; Comprehensive Radiation Therapy
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Adjuvant Hypofractionated Radiation (Experimental): Adjuvant Hypofractionated Radiation (4005 cGy) will last 3-4 weeks with 15 treatments, +/- 4 additional fractions as a boost. Radiation should commence within 180 days of the date of primary surgery. Four additional fractions (a "boost" or "conedown") to areas deemed to be at particularly high risk of recurrence may be added at the end of the radiation course. Fraction size for the boost treatment will continue at 267 cGy for an additional 1068 cGy in four fractions.
  Interventions: Combination Product: Adjuvant Hypofractionated Radiation

INTERVENTIONS:
Combination Product: Adjuvant Hypofractionated Radiation — Hypofractionation is the delivery of radiotherapy in single daily doses greater than the 180-200 cGy. Hypofractionation, through use of larger doses per fraction and fewer total treatments, is a method of shortening overall treatment time in breast cancer therapy.
  Other Names: Radiation Therapy

SUMMARY:
The proposed study is being done to learn more about a particular dose of radiation treatment for breast cancer that is completed in a shorter amount of time than what has traditionally been used to treat breast cancer. Subjects are being asked to be in this research study because they have already had surgery for breast cancer and some cancer cells were found in their lymph nodes that drain the breast tissue.

DETAILED DESCRIPTION:
Subjects who join the study will receive a shortened course of radiation treatment that will last approximately four (4) weeks, instead of the traditional six (6) week course that women have typically received in this situation. The shorter course subjects will receive is designed in a way that it is thought to be equivalent to the longer course. This shorter course has already been shown to be very safe and effective when treating breast cancer in the breast tissue only. However, because cancer cells were found in the lymph nodes that drain their breast, subjects require radiation to a larger area of their chest, armpit, and shoulder than has been completely tested with this experimental dose.

ELIGIBILITY:
Inclusion Criteria:

1. Adult women (≥18 years old) with breast cancer who have undergone surgery for their primary breast tumor (either lumpectomy or mastectomy +/- reconstruction) and are confirmed to have involved lymph nodes on surgical pathology.
2. Patient who have undergone either a total mastectomy or a lumpectomy are eligible.

   Acceptable procedures for assessment of axillary nodal status at the time of surgery include:
   * axillary node dissection;
   * sentinel node biopsy alone; or
   * sentinel node biopsy followed by axillary node dissection.
3. Eligible women include AJCC (American Joint Committee on Cancer) 7th ed. Stage cN0 or cN1 subsequently staged after surgery as Stage pIB (N1mic), pIIA, pIIB, pIIIA, pIIIB, or N3a (10 or more axillary nodes) only: note that ypN0 will also be eligible if pathologic confirmation of nodal involvement was documented prior to neoadjuvant chemotherapy and the patient was found to be node-negative at the time of surgery. Note that women less than 50 years of age, women who received chemotherapy, patients staged as pN0 (i+ or mol+), and large-breasted women are eligible for enrollment.
4. The patient must have recovered from surgery with the incision completely healed and no signs of infection. If adjuvant chemotherapy was administered, chemotherapy-related toxicity that may interfere with delivery of radiation therapy should have resolved. The patient must have an ECOG performance status of 0 or 1 (KPS >70%).
5. The interval between the last surgery for breast cancer (including re-excision of margins) and randomization must be no more than 180 days if chemotherapy is not delivered adjuvantly. If adjuvant chemotherapy was administered, the interval between the last chemotherapy treatment and randomization must be no more than 180 days.
6. Before the patient is enrolled, the consent form, including any addenda, must be signed and dated by the patient and the person who explains the study to that patient.
7. Subjects will have the ability to understand, and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. patients <18 years old
2. pregnant women
3. male patients
4. women with T4 disease, including inflammatory breast cancer
5. women who have declined or otherwise not received preceding surgery
6. women with positive margins after primary surgery
7. women with node-negative disease
8. women without histologic confirmation of nodal involvement
9. women more than 180 days out from primary breast surgery or adjuvant chemotherapy
10. patients with clinically detected or suspicious lymph node involvement not readily amenable to surgical treatment (≥cN2 disease)
11. patients with synchronous bilateral breast cancers
12. patients with prior ipsilateral thoracic or breast radiation
13. patients with distant metastatic disease (cM1) or a life expectancy of less than 5 years
14. active collagen vascular disease, specifically dermatomyositis with a CPK level above normal or with an active skin rash, systemic lupus erythematosus, or scleroderma.
15. other non-malignant systemic disease that would preclude the patient from receiving study treatment or would prevent required follow-up.
16. patients with psychiatric or addictive disorders or other conditions that, in the opinion of the Investigator, would preclude the patient from meeting the study requirements.
17. patients with a separate non-cutaneous cancer diagnosis for which the patient has not been without evidence of disease for at least 5 years.

Note: women <50 years of age, women who received chemotherapy, pN0 (i+ or mol+), and large-breasted women are eligible for enrollment.

Ages: 18 Years to 101 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2016-08-11 (Actual); Primary Completion 2024-06-13 (Actual); Study Completion 2026-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Fisher, MD, MPH, Principal Investigator — University of Colorado, Denver
Locations (3):
- United States (3):
  - University of Colorado Hospital, Aurora, Colorado
  - Memorial Hospital, Colorado Springs, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adjuvant Hypofractionated Radiation
Started | 108
Completed | 63
Not Completed | 45

BASELINE CHARACTERISTICS:
Arm/Group | Adjuvant Hypofractionated Radiation
Number analyzed (Participants) | 108
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53 [46 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 91
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 84
  More than one race | 6
  Unknown or Not Reported | 8
Region of Enrollment [Number; unit: participants]
  United States | 108

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Treatment-related Adverse Event of Interest
Description: The composite endpoint is "yes" for a given patient if that patient experienced at least one of six component adverse events: lymphedema, shoulder ROM impairment, cardiac ischemia, symptomatic rib fracture, brachial plexopathy Grade 2 ('moderate symptoms; limiting instrumental activity of daily living (ADL)') or Grade 3 ('severe symptoms; limiting self-care ADL'), or Grade 2 pneumonitis (requires steroids). AEs were assessed by CTCAE version 4.03.
Time Frame: 12 months and 36 months
Population: Patients are included in analysis for this outcome measure if they have an event recorded for at least one of the six components of the composite endpoint, or if they had non-missing data for all six components.
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Hypofractionated Radiation
Number analyzed (Participants) | 90
Participants
  12 months | 15
  36 months: number analyzed (Participants) | 76
  36 months | 20

2. Primary Outcome: Number of Participants With Lymphedema Severity by Measuring Interlimb Circumference
Description: An increase in interlimb arm circumference of at least 10% in the lower arm or the upper arm, or both, compared with the contralateral arm at the same timepoint, will be judged to be clinically significant lymphedema. Arm circumference 15 cm above the medial epicondyle (upper arms) and 15 cm below the medial epicondyle (lower arms) will be assessed at 12 months and at 36 months.
Time Frame: 12 months and 36 months
Population: Patients who were missing a follow-up assessment at the given dates were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Hypofractionated Radiation
Number analyzed (Participants) | 90
Participants
  12 months | 11
  36 months: number analyzed (Participants) | 77
  36 months | 15

3. Primary Outcome: Number of Participants With Symptomatic Rib Fracture as Measured by Plain Film or CT
Description: Symptomatic rib fracture will be diagnosed by evidence of a correlative lesion on plain film or CT.
Time Frame: 12 months and 36 months
Population: Patients who were missing a follow-up assessment at the given times for this endpoint were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Hypofractionated Radiation
Number analyzed (Participants) | 92
Participants
  12 months | 0
  36 months: number analyzed (Participants) | 74
  36 months | 0

4. Primary Outcome: Number of Participants With New Development of Ischemic Heart Disease as Measured by EKG
Description: Ischemic heart disease will be measured by the new development of angina with corresponding EKG changes, or myocardial infraction.
Time Frame: 12 months and 36 months
Population: Patients who were missing a follow-up assessment for this outcome measure at the given time points were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Hypofractionated Radiation
Number analyzed (Participants) | 92
Participants
  12 months | 0
  36 months: number analyzed (Participants) | 74
  36 months | 0

5. Primary Outcome: Number of Participants Reporting Shoulder Stiffness as Measured by the EORTC QLQ-BR23
Description: Shoulder stiffness severity is assessed using the European Organization for Research and Treatment of Cancer Quality of Life questionnaire breast cancer module (EORTC QLQ-BR23). It is assessed based on patient response to the questionnaire item, "During the past week, was it difficult to raise your arm or to move it sideways?", which is scored from 1 to 4 with 1 being "not at all" and 4 being "very much". Shoulder stiffness is identified in a patient when their response to that question is 3 or 4 AND if their response increased numerically from their response on day 1.
Time Frame: 12 months and 36 months
Population: Patients were excluded if they were missing data for this event.
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Hypofractionated Radiation
Number analyzed (Participants) | 92
Participants
  12 months | 5
  36 months: number analyzed (Participants) | 74
  36 months | 6

6. Primary Outcome: Number of Participants With Grade 2 or Higher Pneumonitis
Description: Number of patients who experience pneumonitis as an adverse event at Grade 2 or higher as assessed by CTCAE v 4.03.
Time Frame: 12 months and 36 months
Population: Patients who were missing an assessment for this endpoint were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Hypofractionated Radiation
Number analyzed (Participants) | 90
Participants
  12 months | 0
  36 months: number analyzed (Participants) | 74
  36 months | 0

7. Primary Outcome: Number of Participants With Grade 2 or Higher Brachial Plexopathy
Description: Number of patients who experience brachial plexopathy as an adverse event at Grade 2 or higher as assessed by CTCAE v 4.03.
Time Frame: 12 months and 36 months
Population: Patients who were missing an assessment for this endpoint were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Hypofractionated Radiation
Number analyzed (Participants) | 92
Participants
  12 months | 0
  36 months: number analyzed (Participants) | 74
  36 months | 0

8. Secondary Outcome: Number of Participants With Disease Recurrence
Description: Recurrent disease presentation within axillary lymph node levels I, II, or III. The supraclavicular region is not included in this endpoint.
Time Frame: Up to 60 months
Population: 2 subjects of 108 total were excluded due to having no follow-up data.
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Hypofractionated Radiation
Number analyzed (Participants) | 106
Participants | 0

9. Secondary Outcome: Number of Participants With Metastasis-free Survival
Description: Measured by the time from date of enrollment to earlier of clinical detection of metastatic disease beyond the breast/chestwall and regional lymph nodes or death.
Time Frame: 12 months and 36 months
Population: 2 participants who did not have a follow-up visit to assess metastasis status were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Hypofractionated Radiation
Number analyzed (Participants) | 106
Participants
  12 months | 106
  36 months | 103

10. Secondary Outcome: Number of Participants With Local-regional Failure Free Survival
Description: Measured by the time from date of enrollment to earlier of clinical detection of any ipsilateral recurrent disease to the breast/chestwall or regional lymph nodes (levels I, II, III, supraclavicular, and internal mammary lymph nodes) or death.
Time Frame: 12 months and 36 months
Population: 2 participants did not have a follow-up visit where local or regional disease recurrence was assessed and were excluded from this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Hypofractionated Radiation
Number analyzed (Participants) | 106
Participants
  12 months | 106
  36 months | 104

11. Secondary Outcome: Number of Participants With a Change in Quality of Life Score as Measured by the EORTC QLQ-C30
Description: Patient's quality of life from pre-treatment to post-treatment, reported by the quality of life questionnaire [EORTC QLQ-C30 V1]. Summary scores and missing data handling were performed according to the EORTC QLQ-C30. The minimum score is 0, and the maximum score is 100. A higher score is a better outcome. A change in score is defined as a score increase of at least 10 points at the 12 month mark compared to baseline.
Time Frame: From baseline up to 12 months
Population: This is the number of patients who completed the EORTC QLQ-C30 at both baseline and 1 year post-intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Hypofractionated Radiation
Number analyzed (Participants) | 86
Participants | 21

12. Secondary Outcome: Number of Participants With a Change in Quality of Life Score as Measured by the EORTC QLQ-BR23
Description: Patient's quality of life from pre-treatment to post-treatment, reported by the quality of life questionnaire breast cancer module [EORTC QLQ-BR23 V1]. Summary scores and missing data handling were performed according to the EORTC QLQ-BR23. The minimum score is 0, and the maximum score is 100. A higher score is a better outcome. A change in score is defined as a score increase of at least 10 points from baseline.
Time Frame: Baseline to 1 year post-intervention
Population: This is the number of patients who completed the EORTC QLQ-BR23 at both baseline and 1 year post-intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Hypofractionated Radiation
Number analyzed (Participants) | 79
Participants | 17

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Adjuvant Hypofractionated Radiation
All-Cause Mortality (participants affected / at risk) | 6/108
Serious Adverse Events (participants affected / at risk) | 11/108
Other Adverse Events (participants affected / at risk) | 108/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adjuvant Hypofractionated Radiation (N=108)
Skin infection (Infections and infestations) | 1 (2) — Cellulitis
Breast infection (Infections and infestations) | 1 (1)
Brain mets/progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Death NOS (General disorders) | 2 (2)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adjuvant Hypofractionated Radiation (N=108)
Fatigue (General disorders) | 70
Dysphagia (Gastrointestinal disorders) | 45
Breast pain (Reproductive system and breast disorders) | 34
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 34
Hot flashes (Vascular disorders) | 30
Erythema (Skin and subcutaneous tissue disorders) | 56
Pruritis (Skin and subcutaneous tissue disorders) | 22 — Simply recorded as pruritis.
Lymphedema (Vascular disorders) | 19
Nausea (Gastrointestinal disorders) | 17
Dermatitis (Skin and subcutaneous tissue disorders) | 15
Dermatitis radiation (Injury, poisoning and procedural complications) | 22
Esophagitis (Gastrointestinal disorders) | 14
Sore throat (Respiratory, thoracic and mediastinal disorders) | 12
Anxiety (Psychiatric disorders) | 11
Insomnia (Psychiatric disorders) | 10
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Neuropathy (Nervous system disorders) | 9
Breast tenderness (General disorders) | 8
Headache (Nervous system disorders) | 13
Vaginal dryness (Reproductive system and breast disorders) | 8
Desquamation (Skin and subcutaneous tissue disorders) | 7
Chest tightness (Cardiac disorders) | 6
Chest wall pain (Musculoskeletal and connective tissue disorders) | 6
Constipation (Gastrointestinal disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-10-08): https://cdn.clinicaltrials.gov/large-docs/86/NCT02700386/Prot_SAP_ICF_000.pdf